CLINICAL TRIAL: NCT00898885
Title: Clinical and Histological Evaluation of Chronic Graft-Versus Host Disease (cGVHD) in Oral Mucosa
Brief Title: Analysis of the Clinical and Histological Correlation of Oral Graft-Versus-Host-Disease (GVHD)
Acronym: ORALGVHD
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Paulo Sérgio da Silva Santos, School of Dentistry - Oral Pathology
Other Study IDs: OPPSSS1
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Graft-Versus-Host Disease
Keywords: oral manifestations; bone marrow transplantation; adverse effects
MeSH Terms: conditions — Graft vs Host Disease; Oral Manifestations | interventions — Biopsy; Bone Marrow Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples of oral mucosa and minor salivary glands stained with hematoxylin and eosin for visualization of the layers in optical microscope
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Bone Marrow Transplantation
  Interventions: Procedure: oral biopsy

INTERVENTIONS:
Procedure: oral biopsy — oral mucosa and salivary gland biopsy after bone marrow transplantation
  Other Names: oral manifestations; graft-versus-host disease; bone marrow transplantation

SUMMARY:
Introduction: Graft-versus-host-disease (GVHD) is the major cause of morbidity and mortality in patients submitted to the Bone Marrow Transplantation (BMT). The oral manifestations can be very debilitating and interfere in the results of medical therapy, leading to systemic complications, committing the prognosis and quality of life of the patient.

The early diagnosis can be done through biopsies of oral mucosa with or without apparent injury clinic. The association between the clinical and histopathological tables of GVHD, especially through the use of recent consensus established in these areas, can bring new benefits to physicians.

Objective: This study aims to apply and compare the two classifications histological to GVHD, Horn (1995) and Consensus (2006) in specimens obtained from clinical oral lesions suggestive of GVHD; correlate them with clinical classification according Akpek (2001) and with the survival of the patients.

DETAILED DESCRIPTION:
Methods: For this study we analyzed histological samples of oral mucosa of 10 patients with clinical diagnosis of GVHD, which have areas of epithelium, and salivary gland. The histopathological aspects were observed by the author of this work and his advisor, so blinded by applying the criteria for Horn and the Consensus. We consistency between the two classifications obtained and histological correlation with the clinical classification of GVHD (Akpek, 2001) and the curve of survival.

ELIGIBILITY:
Inclusion Criteria:

* all patients with clinical signs of oral GVHD that underwent oral biopsy

Exclusion Criteria:

* samples without epithelium or minor salivary glands

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients underwent bone marrow transplantation with clinical signs of oral Graft-versus-host Disease
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The histological classification according Horn showed that in most cases there was presence of GVHD with low degrees of severity; Already classification of the Consensus showed that there were in full presence of GVHD of moderate degree. | during the survey data, and analysis of specimens

CONTACTS AND LOCATIONS:
Overall Officials: Marina HG Magalhães, DMD, PhD, Study Chair — University of Sao Paulo - Brazil